CLINICAL TRIAL: NCT05564624
Title: A Clinical Study to Determine the Facial Skin Benefits of a Periodic Fasting-Mimicking Diet
Brief Title: Effect of Fasting-Mimicking Diet on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L-Nutra Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LNT21-006; C21-D192 (Other: SGS Stephens, Inc)
Record Dates: First submitted 2022-09-18; First posted 2022-10-03 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Skin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No usage instructions. Continue regular eating habits for the duration of the study.
- Fasting Mimicking Diet (Experimental): Use the test products, ProLon(TM) Fasting Mimicking Diet, during the scheduled 5-day period in place of the usual meals (breakfast, lunch, dinner, snack) according to the instructions. Use the test product for 5 days for 3 cycles, beginning on day 1, day 30, and day 60.
  Interventions: Other: Fasting mimicking diet (FMD)

INTERVENTIONS:
Other: Fasting mimicking diet (FMD) — The ProLon(TM) Fasting Mimicking Diet regimen is a meal replacement plan that mimics water only fasting. It consists of 100% natural ingredients, which are generally regarded as safe (GRAS). It is comprised of bars, soups, and beverages aiming to achieve consistent and effective short-term calorie restriction, while providing adequate micronutrients. The very low protein and very low sugar content are essential characteristics of the diet. Complex carbohydrates and polyunsaturated fatty acids are its main components.
  Arms: Fasting Mimicking Diet

SUMMARY:
This single-center, randomized, controlled clinical trial is being conducted to assess the efficacy on facial skin appearance of the Sponsor's 5-day meal kit when consumed monthly for 3 cycles over the course of 71 days by women with mild to moderate dry fine lines, lack of smoothness, uneven skin tone, and lack of radiance on the face.

DETAILED DESCRIPTION:
Fasting-mimicking diet (FMD) was developed to mimic the metabolic effects of water-only fasting, while providing modest calories and essential nutrients. It consists of 100% natural ingredients, which are generally regarded as safe (GRAS). It is comprised of bars, soups, and beverages aiming to achieve consistent and effective short-term calorie restriction, while providing adequate micronutrients.

The study will test the efficacy parameters, including clinical grading scores, Corneometer measurement, and Antera image analysis and subject self-assessment, of consuming the test products in place of other food over a 5 day period, for 3 cycles, over the course of 71 days when compared with baseline scores/values, and when compared to the untreated control.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 35 to 60 years of age.
2. In good general health (physical, mental, and social well-being, not merely the absence of disease/infirmity), according to subject self-report.
3. Having mild to moderate (score of 3-6 according to a modified Griffiths scale,11 where 0=none and 9=severe) scores for the following parameters on the global face: Dry fine lines, Roughness/skin smoothness (visual), Uneven skin tone, Dullness/lack of radiance
4. Having a Body Mass Index in the range of 20-35 at the baseline visit.
5. Having not had any facial treatments in the past 6 months and are willing to withhold all facial treatments during the course of the study including facials, facial peels, photo facials, laser treatments, dermabrasion, botulinum toxin (Botox®), injectable filler treatments, intense pulsed light (IPL), acid treatments, tightening treatments, facial plastic surgery, or any other treatment administered by a physician or skin care professional designed to improve the appearance or firmness of facial skin. Waxing and threading are allowed but not facial laser hair removal.

Exclusion Criteria:

1. Having known allergy or sensitivity to food or any component of the meal kit, including nuts, celeriac/celery, oats, and sesame. (Some of the products [bars] are processed in a facility where peanuts, eggs, soy, wheat, milk, and shellfish are also present.)
2. Breastfeeding, pregnant, or planning to become pregnant during the study according to subject self-report.
3. Having fasted (abstained from food) or having followed a very restricted food plan (eg, a cleanse or fast mimicking diet)for any period of more than 24 hours in the past 90 days.
4. Having a history of gastric bypass.
5. Having or having a history of a known, suspected, or diagnosed condition of disordered or restricted eating.
6. Currently experiencing menopause or having experienced menopause within the last 12 months. 9. Having a history of skin cancer within the past 5 years.
7. Having a health condition and/or pre-existing or dormant dermatologic disease on the test area/face that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
8. Having observable sunburn, suntan, scars, nevi, excessive hair, tattoos, or other dermal conditions on the test areas that might influence the test results in the opinion of the Investigator or designee.
9. Having a history of immunosuppression/immune deficiency disorders, organ transplant, or currently using oral or systemic immunosuppressive medications and biologics and/or undergoing radiation or chemotherapy as determined by study documentation.
10. Currently using or having regularly used corticosteroids (systemic or topical, not nasal or ocular) within the past 4 weeks.
11. Having or having a history of diabetes, epilepsy, liver failure, advanced chronic kidney disease, heart failure, or syncope (fainting), or other metabolic disorder or serious health condition.
12. Having a risk for recurrent infections or currently experiencing a fever, cough, diarrhea, or active yeast infection.
13. Having a disease such as asthma, hypertension, hyperthyroidism, or hypothyroidism that is not controlled by diet or medication, or hypertension requiring treatment with more than one medication. Individuals having multiple or severe health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
14. Having started a long-term medication within the last 2 months.
15. Having any planned surgeries or invasive medical procedures during the study (including colonoscopy). Noninvasive medical procedures or surgeries will be reviewed for their impact on the study outcome and acceptability by the Investigator or designee.
16. Currently participating in any other clinical trial.
17. Having participated in any clinical trial involving the face within 2 weeks before study enrollment.
18. Having started hormone replacement therapies (HRT) or hormones for birth control or menopause less than 3 months before study enrollment or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
19. Has any medical disease or condition that, in the opinion of the principal investigator (PI) or appropriate study personnel, precludes study participation.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical grading of the facial skin | Day 0 (baseline) and 71
  Clinical grading will be assessed on the indicated location on each subject's face using a modified Griffiths 10-point scale according to the following numerical definitions. Half-point scores may be used as necessary to more accurately describe the skin condition:
  1. Skin smoothness (visual), cheeks;
  2. Skin smoothness (tactile), cheeks;
  3. Dry fine lines, global face;
  4. Clarity, global face;
  5. Redness, global face;
  6. Evenness of skin tone, global face;
  7. Radiance, global face;
  8. Overall appearance of skin condition (health)

SECONDARY OUTCOMES:
Clinical grading of the facial skin | Day 0 (baseline) and day 11
  Clinical grading will be assessed on the indicated location on each subject's face using a modified Griffiths 10-point scale according to the following numerical definitions. Half-point scores may be used as necessary to more accurately describe the skin condition:
  1. Skin smoothness (visual), cheeks;
  2. Skin smoothness (tactile), cheeks;
  3. Dry fine lines, global face;
  4. Clarity, global face;
  5. Redness, global face;
  6. Evenness of skin tone, global face;
  7. Radiance, global face;
  8. Overall appearance of skin condition (health)
Facial skin hydration | Day 0 (baseline) and day 11
  Triplicate Corneometer (Corneometer CM 825, Courage + Khazaka electronic GmbH, Köln, Germany) measurements will be taken on the center of each subject's right cheek (at the intersection of lines extending up from the corner of the mouth and horizontally across the bottom of the nose). The Corneometer measures moisture content in the stratum corneum by an electrical capacitance method. The measurement has no units, but is proportional to the dielectric constant of the surface layers of the skin, and increases as the skin becomes more hydrated. The readings are directly related to the skin's electrical capacitance (picofarads).
Facial skin hydration | Day 0 (baseline) and day 71
  Triplicate Corneometer (Corneometer CM 825, Courage + Khazaka electronic GmbH, Köln, Germany) measurements will be taken on the center of each subject's right cheek (at the intersection of lines extending up from the corner of the mouth and horizontally across the bottom of the nose). The Corneometer measures moisture content in the stratum corneum by an electrical capacitance method. The measurement has no units, but is proportional to the dielectric constant of the surface layers of the skin, and increases as the skin becomes more hydrated. The readings are directly related to the skin's electrical capacitance (picofarads).
Digital Imaging by VISIA | Day 0 (baseline) and day 11
  VISIA-CR Imaging (Canfield Imaging Systems, Fairfield, New Jersey) with a Canon Mark II digital SLR camera (Canon Incorporated, Tokyo, Japan).
Digital Imaging by VISIA | Day 0 (baseline) and day 71
  VISIA-CR Imaging (Canfield Imaging Systems, Fairfield, New Jersey) with a Canon Mark II digital SLR camera (Canon Incorporated, Tokyo, Japan).
Digital Imaging | Day 0 (baseline) and day 11
  Digital Imaging Using Portrait Photo Station (Canon Mark II 7D digital SLR camera (Canon Incorporated, Tokyo, Japan) with a Canon EF-S 60mm f/2.8 macro lens with visible lighting mode.).
Digital Imaging | Day 0 (baseline) and day 71
  Digital Imaging Using Portrait Photo Station (Canon Mark II 7D digital SLR camera (Canon Incorporated, Tokyo, Japan) with a Canon EF-S 60mm f/2.8 macro lens with visible lighting mode.).
Digital Imaging for skin roughness | Day 0 (baseline) and day 11
  Antera 3D Imaging (Miravex Ltd, Dublin, Ireland).
Digital Imaging for skin roughness | Day 0 (baseline) and day 71
  Antera 3D Imaging Procedures (Miravex Ltd, Dublin, Ireland).
Self-assessment | Day 0 (baseline) and day 11
  Skin condition self-assessment questionnaire
Self-assessment | Day 0 (baseline) and day 71
  Skin condition self-assessment questionnaire on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Summer Acevedo, PhD, Principal Investigator — SGS Stephens, Inc
Locations (1):
- SGS Stephens, Inc, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No